CLINICAL TRIAL: NCT02583425
Title: Pilot Study of DFN-11 Injection in Medication Overuse Headache
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFN-11-CD-007
Record Dates: First submitted 2015-10-01; First posted 2015-10-22 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-02

CONDITIONS: Medication Overuse Headache
MeSH Terms: conditions — Headache Disorders, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DFN-11 (Experimental): DFN-11 Injection upon occurrence of migraine
  Interventions: Drug: DFN-11 Injection

INTERVENTIONS:
Drug: DFN-11 Injection

SUMMARY:
Efficacy and Safety Pilot Study of DFN-11 Injection in Medication Overuse Headache

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of medication overuse headache within the past year in the following categories
2. Diagnosis of migraine, with or without aura for at least 12 months
3. Experience an average of > 10 headache days per month for the past 12 months
4. Females must:

   i. be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method [e.g., condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel], or male partner sterilization) before entry and willing to continue throughout the study, or ii. be surgically sterile, (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), or iii. be postmenopausal (spontaneous amenorrhea for at least 1 year)
5. Females of child-bearing potential must have a negative urine pregnancy test at all visits.
6. Able and willing to read and comprehend written instructions and complete the electronic diary.
7. Must have internet access to complete daily headache diary.

Exclusion Criteria:

1. Current use of medication for headache/migraine prophylaxis that has not been stable for 30 days prior to screening. Stable is defined as no recent dosing change within 30 days of screening.
2. Hemiplegic or basilar migraine
3. History, symptoms or signs of ischemic cardiac, cerebrovascular or peripheral vascular syndromes
4. Uncontrolled hypertension (screening systolic/diastolic blood pressure > 140/90 mmHg in 2 out of 3 readings)
5. Clinically significant hepatic impairment
6. History of epilepsy or conditions associated, which in the opinion of the Investigator, increase the likelihood of present day seizure
7. History (within 2 years) of drug or alcohol abuse as defined by DSM-IV-TR criteria
8. Systemic disease, which in the opinion of the Investigator, would contraindicate participation
9. History of a neurological or psychiatric condition, which in the opinion of the Investigator would contraindicate participation
10. Pregnant or lactating women
11. Have taken any investigational medication within 30 days before screening, or are scheduled to receive an investigational drug
12. Subjects with a positive urine drug screen for recreational drugs or marijuana (whether legal or not) or for prescription drugs not explained by stated concomitant medications
13. Clinical laboratory or electrocardiogram (ECG) abnormality that in the opinion of the Investigator would endanger the subject or interfere with the study conduct. If the results of the clinical laboratory or ECG are outside of normal reference range the subject may still be enrolled but only if these findings are determined to be not clinically significant by the Investigator. This determination must be recorded in the subject's source document prior to enrolment.
14. Fridericia's corrected QT (QTcF) interval greater than 450 msec
15. Severe renal impairment (creatinine > 2 mg/dl)
16. Serum total bilirubin > 2.0 mg/dL
17. Serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase > 2.5 times the upper limit of normal
18. Subjects with uncontrolled diabetes mellitus, or a glycosylated hemoglobin (HbA1c) > 7.0%, or with diabetes mellitus requiring insulin
19. Subjects who in the opinion of the investigator experience rebound headache from caffeine usage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinvest, Springfield, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Screening
Arm/Group | DFN-11
Started | 27
Completed | 15
Not Completed | 12
Not completed — Did not meet entry criteria | 12
Period: Baseline
Arm/Group | DFN-11
Started | 15
Completed | 10
Not Completed | 5
Not completed — Did not meet continued criteria | 5
Period: Treatment Period
Arm/Group | DFN-11
Started | 10
Completed | 9
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | DFN-11
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Headache Hours in the Baseline Period (28 Days of Subjects Using Their Usual Medication for Headaches) and in the Treatment Period (28 Days of Subjects Using DFN-11 for Headaches)
Time Frame: 28 days Baseline period and 28 days of Treatment period (Total 56 days)
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- DFN-11: DFN-11 Injection upon occurrence of migraine headache
  DFN-11 Injection
Arm/Group | DFN-11
Number analyzed (Participants) | 9
Hours
  Baseline period | 202.82 (152.58)
  Treatment period | 138.71 (113.60)

2. Secondary Outcome: The Number of Acute Headache Medication Doses in the Baseline Period (28 Days of Subjects Using Their Usual Medication for Headaches) and in the Treatment Period (28 Days of Subjects Using DFN-11 for Headaches)
Time Frame: 28 days Baseline period and 28 days of Treatment period (Total 56 days)
Measure: Mean (Standard Deviation); unit: Number of doses of acute medication used
Groups:
- DFN-11: DFN-11 Injection upon occurrence of migraine
  DFN-11 Injection
Arm/Group | DFN-11
Number analyzed (Participants) | 9
Number of doses of acute medication used
  Baseline period | 16.56 (3.43)
  Treatment period | 19.78 (10.13)

ADVERSE EVENTS:
Arm/Group | DFN-11
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFN-11 (N=10)
Dsypepsia (Gastrointestinal disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Arthralgia (General disorders) | 1 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No